CLINICAL TRIAL: NCT00215150
Title: Ziprasidone for the Treatment of Refractory Social Anxiety Disorder
Brief Title: Geodon for the Treatment of Refractory Social Anxiety Disorder
Acronym: SAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00012882; 6479 (Other: Duke legacy protocol number)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2013-05-24 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2013-04

CONDITIONS: Social Anxiety Disorder
Keywords: anxiety disorder; SAD; ziprasidone; sertraline; antidepressant; antipsychotic
MeSH Terms: conditions — Phobia, Social; Anxiety Disorders | interventions — ziprasidone; Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Open Label Treatment (Other): 8 weeks of open label treatment with sertraline
  Interventions: Drug: Sertraline
- Randomization Ziprasidone (Other): 8 weeks of treatment with sertraline augmented with ziprasidone
  Interventions: Drug: Ziprasidone; Drug: Sertraline
- Randomization Placebo (Other): 8 weeks of treatment with sertraline augmented by placebo
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Ziprasidone — Sertraline augmentation with ziprasidone
  Other Names: Geodon
  Arms: Randomization Ziprasidone
Drug: Sertraline — Treatment by sertraline in open label phase, followed by ziprasidone/placebo randomized augmentation in the randomized phase
  Other Names: Zoloft

SUMMARY:
The purpose of this study is to examine the effectiveness and tolerability of augmentation treatment of ziprasidone to achieve remission among patients with social anxiety disorder (SAD) who did not remit on sertraline treatment alone

DETAILED DESCRIPTION:
This is a two-phase study consisting of 8 weeks of open label treatment with sertraline (50-200 mg/day) in patients with SAD and in those who fail to demonstrate symptom remission on sertraline alone, 8 weeks of randomized, double-blind, placebo-controlled augmentation with ziprasidone.

ELIGIBILITY:
Inclusion Criteria:

* adults 18-65 years of age
* primary diagnosis of SAD, using Diagnostic Standard Manual(DSM-IV) criteria
* minimum Clinical Global Impression of Severity (CGI-S) score of 4 at baseline
* minimum Brief Social Phobia Scale(BSPS) score of 20 at baseline
* written informed consent
* negative serum pregnancy test for women of childbearing potential
* normal EKG

Exclusion Criteria:

* current DSM-IV diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, mental retardation or other pervasive developmental disorder, or cognitive disorder due to a general medical condition
* any current primary anxiety disorder other than SAD
* current primary depression
* history of substance abuse or dependence within the last 3 months
* suicide risk or serious suicide attempt within the last year
* clinically significant medical condition or laboratory or EKG abnormality
* women of childbearing potential who are unwilling to practice an acceptable method of contraception
* patients needing concurrent use of psychotropic medications
* history of hypersensitivity to sertraline or ziprasidone
* recent (less than 2 months) initiation of psychotherapy for SAD
* history of failure to respond to augmentation with an adequate trial of an atypical antipsychotic
* patients who are currently taking any of the following medications: Erythromycin, Biaxin, Avelox, Zithromax, Amantadine, Levaquin, Tamoxifen, Tegretol, Nizoral, and Levitra

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-11; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Davidson JR, Potts NL, Richichi EA, Ford SM, Krishnan KR, Smith RD, Wilson W. The Brief Social Phobia Scale. J Clin Psychiatry. 1991 Nov;52 Suppl:48-51. doi: 10.1037/t07672-000. PMID 1757457

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from the immediate surrounding area, by use of Institutional Review Board (IRB) approved television and radio advertisements, along with flyers.
Groups:
- Open Label Treatment: 8 weeks of open label treatment with sertraline (50-200mg/day)followed by 8 weeks of randomized, Double Blind (DB), placebo-controlled augmentation with ziprasidone (40-160mg/day)for qualifying subjects.
Period: Open Label Phase
Arm/Group | Open Label Treatment
Started | 51 (Number of subjects consented)
Completed | 21
Not Completed | 30
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 1
Not completed — Did not complete a post base visit | 13
Not completed — Did not meet randomization criteria | 9
Period: Randomization Phase Ziprasidone
Arm/Group | Open Label Treatment
Started | 10
Completed | 7
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Period: Randomization Phase Placebo
Arm/Group | Open Label Treatment
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: This is the intent to treat population consisting of subjects completing at least one post baseline visit.
Groups:
- Study Treatment: 8 weeks of open label treatment with sertraline followed by 8 weeks of treatment with ziprasidone/placebo for qualifying subjects
Arm/Group | Study Treatment
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Brief Social Phobia Scale(BSPS)
Description: An observer measure of social phobic symptoms, referred to as the Brief Social Phobia Scale, consists of 11 items, 7 evaluating commonly feared or avoided situations and 4 additional items measuring autonomic distress. A total numerical range of 0-88 is scored on this measure, with higher scores representing greater severity of social anxiety disorder symptoms.The total score is computed as a simple sum of the 11 items.
Time Frame: Baseline, 8 and 16 weeks
Population: The number of participants evaluated in either phase is based on a last observation carried forward analysis requiring at least one visit completed in addition to the first timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open Label Phase: The open label treatment phase for the first 8 weeks
- Randomization Phase for Ziprasidone Group: The group of subjects randomized to receive Ziprasidone for the second 8 weeks
- Randomization Phase for Placebo Group: The group of subjects randomized to receive placebo for the second 8 weeks
Arm/Group | Open Label Phase | Randomization Phase for Ziprasidone Group | Randomization Phase for Placebo Group
Number analyzed (Participants) | 38 | 10 | 11
units on a scale
  Beginning of Study Phase | 44.0 (11.1) [24 to 67] | 31.8 (8.9) [18 to 47] | 31.8 (11.8) [12 to 55]
  End of Study Phase | 31.2 (16.0) | 21.0 (13.6) | 24.6 (12.3)
Statistical Analysis 1: Comparison: Open Label Phase; Results are from a Wilcoxon signed rank test on the difference from endpoint to baseline for the intent to treat sample from the open label phase of the project; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Randomization Phase for Ziprasidone Group vs Randomization Phase for Placebo Group; Results are from a Kruskal Wallis test on the ziprasidone/placebo groups from the randomization phase of the project; Test type: Superiority or Other; p > .05, Kruskal-Wallis

ADVERSE EVENTS:
Groups:
- Open Label Phase: The first 8 weeks of treatment on sertraline
- Randomization Phase for Ziprasidone: The second phase of treatment with subjects randomized to ziprasidone augmentation.
- Randomization Phase for Placebo: The second phase of treatment with subjects randomized to placebo augmentation.
Arm/Group | Open Label Phase | Randomization Phase for Ziprasidone | Randomization Phase for Placebo
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/38 | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No